CLINICAL TRIAL: NCT06813105
Title: Exploratory Analysis of Pain and Function Improvement After Radial Pressure Wave Therapy in Plantar Fasciitis.
Brief Title: Outcome After Radial Pressure Wave Therapy in Plantar Fasciitis.
Acronym: RPWT
Status: Completed | Type: Observational
Sponsor: Hospital Civil de Guadalajara (Other)
Collaborators: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Armando Tonatiuh Avila Garcia, Chief Department of Physical Medicine and Rehabilitation, Hospital Civil de Guadalajara
Other Study IDs: CEI 255/24
Record Dates: First submitted 2025-01-24; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Fasciitis, Plantar; Fasciitis, Plantar, Chronic
Keywords: plantar fasciitis; rehabilitation outcomes
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore potential associations between baseline patient characteristics (such as age, body mass index, and baseline pain intensity) and clinical outcomes in patients with plantar fasciitis undergoing radial pressure wave therapy (RPWT). The study includes male and female adults aged 18 to 60 years.

DETAILED DESCRIPTION:
Background: Plantar fasciitis (PF) is a common cause of heel pain, significantly impairing functionality and quality of life. Radial pressure wave therapy (RPWT) has emerged as a non-invasive therapeutic option. However, there is limited evidence regarding factors that may influence clinical outcomes in patients receiving this treatment.

Objectives: The primary objective of this study is to explore potential associations between baseline patient characteristics (such as age, body mass index, and pain intensity) and clinical outcomes in patients with PF treated with RPWT. Additionally, this study aims to assess changes in pain intensity and functionality following RPWT.

Materials and Methods: This is an exploratory, pilot observational study including patients diagnosed with PF who undergo three sessions of RPWT. The study evaluates changes in pain intensity, assessed using the Numerical Pain Rating Scale (NPRS), and functionality, measured using the WHODAS 2.0. Patient characteristics such as age, body mass index (BMI), and PF chronicity are collected retrospectively from medical records. Statistical analyses will be conducted to examine potential associations between patient characteristics and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plantar fasciitis confirmed by clinical evaluation.
* Age 18 to 60 years.
* Symptoms persisting for at least three months before treatment.
* Completed three RPWT sessions using a standardized protocol (2000 impulses per session, 10 Hz, and 3.5 bar).
* Availability of complete medical records, including three-month follow-up data.

Exclusion Criteria:

* History of foot surgery or corticosteroid injection in the affected limb within the past six months.
* Pregnancy at the time of treatment.
* Presence of concurrent musculoskeletal conditions (e.g., fractures, active infections, sprains) in the affected limb.
* Diagnosis of systemic conditions (e.g., cancer, osteoporosis, autoimmune diseases).
* Incomplete medical records or failure to complete RPWT sessions and follow-up visits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study focuses on adult patients diagnosed with plantar fasciitis (PF), a condition commonly affecting middle-aged individuals. Eligible participants are between 18 and 60 years old and present with symptoms persisting for at least three months before treatment. Given that risk factors such as body mass index (BMI) and physical activity levels may influence clinical outcomes, these characteristics will be documented for all participants. Additionally, data on prior conventional physical therapy and PF chronicity (acute vs. chronic cases) will be collected to explore potential associations with treatment response.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessed by the Numerical Pain Rating Scale (NPRS). | Immediately after the last RPWT session, approximately 1 week after baseline.
  Pain intensity will be measured using the Numerical Pain Rating Scale (NPRS), a validated 10-point scale where 0 represents "no pain" and 10 represents "the worst pain imaginable."

SECONDARY OUTCOMES:
Functionality assessed by the WHODAS 2.0 scale. | Immediately after the last RPWT session, approximately 1 week after baseline.
  Functionality will be evaluated using the WHODAS 2.0, a 12-item questionnaire assessing six domains of disability (cognition, mobility, self-care, interpersonal relationships, life activities, and community participation). Each item is rated on a 5-point scale, where higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: ARMANDO TONATIUH AVILA GARCIA, MD, Principal Investigator — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Charles R, Fang L, Zhu R, Wang J. The effectiveness of shockwave therapy on patellar tendinopathy, Achilles tendinopathy, and plantar fasciitis: a systematic review and meta-analysis. Front Immunol. 2023 Aug 16;14:1193835. doi: 10.3389/fimmu.2023.1193835. eCollection 2023. PMID 37662911
- [Background] Melese H, Alamer A, Getie K, Nigussie F, Ayhualem S. Extracorporeal shock wave therapy on pain and foot functions in subjects with chronic plantar fasciitis: systematic review of randomized controlled trials. Disabil Rehabil. 2022 Sep;44(18):5007-5014. doi: 10.1080/09638288.2021.1928775. Epub 2021 May 26. PMID 34038642
- [Background] Li H, Xiong Y, Zhou W, Liu Y, Liu J, Xue H, Hu L, Panayi AC, Mi B, Liu G. Shock-wave therapy improved outcome with plantar fasciitis: a meta-analysis of randomized controlled trials. Arch Orthop Trauma Surg. 2019 Dec;139(12):1763-1770. doi: 10.1007/s00402-019-03262-z. Epub 2019 Aug 21. PMID 31435724
- [Background] Vahdatpour B, Sajadieh S, Bateni V, Karami M, Sajjadieh H. Extracorporeal shock wave therapy in patients with plantar fasciitis. A randomized, placebo-controlled trial with ultrasonographic and subjective outcome assessments. J Res Med Sci. 2012 Sep;17(9):834-8. PMID 23826009